CLINICAL TRIAL: NCT03639909
Title: Analysis of the Sweat Response According to the Pathology in Neurologic
Brief Title: Analysis of the Sweat Response According to the Pathology in Neurologic Patients
Acronym: Sudoscan
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/15/7550
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Neurological Disorder
Keywords: sweat gland
MeSH Terms: conditions — Nervous System Diseases | interventions — Sweating; Cardiovascular Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MSA-P: Patients with multiple systeme atrophy (MSA) with predominant parkinsonism (MSA-P) had evaluation of cardiovascular function and sweating function
  Interventions: Procedure: sweating function; Procedure: Cardiovascular function
- PD patients: Parkinson's disease (PD) patients had evaluation of cardiovascular function and sweating function
  Interventions: Procedure: sweating function; Procedure: Cardiovascular function

INTERVENTIONS:
Procedure: sweating function — Sweating dysfunction by Sudoscan
  Other Names: sweating dysfunction by Sudoscan
Procedure: Cardiovascular function — Cardiovascular (CV) tests

SUMMARY:
Cardiovascular autonomic neuropathy (CAN) has been shown to be an important risk factor for cardiac diseases, particularly in diabetes.

CAN may be investigated by a battery of laboratory cardiovascular autonomic reflex tests(initially described by Ewing).

First screening for CAN (as proposed in diabetic patients) can be performed by assessing heart rate (HR) response to deep breathing, blood pressure (BP) and HR response to a 5 minutes stand test

DETAILED DESCRIPTION:
Sweat glands are innervated by thin and un myelinated sympathetic C-fibers that can be impaired in neuropathies,especially length-dependent ones. Sweating dysfunction has been shown in several neurological peripheral disorders and it has been suggested that sweating function should be included among the diagnostic tests for the early detection of autonomic neuropathies. Several methods have been developed, but the lack of easy and quick tests to diagnose sweating dysfunction has restricted widespread use in clinical practice. Measurement of electrochemical skin conductance (ESC) using Sudoscan® is a new method for quick, non-invasive and quantitative assessment of sweating. This technique has demonstrated its usefulness in detecting autonomic and small fiber neuropathy, especially in diabetic patients.The aim of this study was to evaluate the performance of the laboratory battery of CV tests and of sweating dysfunction by Sudoscan®, alone or in combination, to differentiate MSA-P from PD. Among the CV tests, the present study particularly looked at those tests already recommended as screening bedside tests in diabetic patients (HR variations with deep breathing and BP variations during stand test) ; these tests are rapid and easy to perform. HR variations with deep breathing depend on parasympathetic tone and BP variations depend on vasomotor sympathetic response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MSA-P or PD

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the autonomic laboratory of the neurology department at Toulouse University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Sweating autonomic test | baseline
  Evaluate the performance of the laboratory battery of CV tests and of sweating dysfunction to differentiate MSA-P from PD

CONTACTS AND LOCATIONS:
Overall Officials: Anne Pavy-Le Traon, MD, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No